CLINICAL TRIAL: NCT01542554
Title: Effect of Low Glycaemic Index Diet on Blood Glucose Control in Chinese Type 2 Diabetic Patients: Randomized Controlled Trial
Brief Title: Effect of Low Glycaemic Index Diet on Blood Glucose Control in Chinese Type 2 Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Ace Lee, Doctor, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKEC-2011-080
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; Chinese; Glycaemic index
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low glycaemic index diet (Experimental)
  Interventions: Other: Low glycaemic index diet
- Usual diabetic diet (Active Comparator)
  Interventions: Other: Usual diabetic diet

INTERVENTIONS:
Other: Low glycaemic index diet — Diabetic subjects will be given dietary advice with emphasis on low glycaemic index diet
  Arms: Low glycaemic index diet
Other: Usual diabetic diet — Diabetic subjects will be given dietary advice without mention about glycaemic index
  Arms: Usual diabetic diet

SUMMARY:
The purpose of this study is to investigate the effect of low glycaemic diet on blood glucose control in Chinese type 2 diabetic patients.

DETAILED DESCRIPTION:
Glycaemic index (GI) is the measurement of post-meal blood glucose rise cause by ingestion of carbohydrate. For the same amount of carbohydrate, food with lower GI value cause a lower post- meal rise in blood glucose concentration in both normal and diabetic patients. Meta-analysis of randomized controlled trial has showed that low GI diet can achieve an additional reduction of A1c by 0.4% when compare with usual diabetic diet. Furthermore, various diabetes associations have already endorsed the use of low GI diet in the management of diabetes.

Hong Kong Chinese obtain most of their carbohydrate intake through consumption of rice or rice related foods, which are considered as having high GI value. In addition, it has been demonstrated that Asian have higher post-prandial rise in blood glucose than Caucasian after consuming the same amount of carbohydrate. When the above two factors add together, we expect our local type 2 diabetic patients are suffering from significant post-prandial hyperglycaemia, which in turn translate into elevated 24-hour hyperglycaemia and A1c.

However, nearly all studies about glycaemic index and diabetes are conducted in Caucasian. It is unclear about the benefit in Chinese patients with type 2 diabetes who are currently having diet with high GI value.

We therefore hypothesized that low GI diet may improve blood glucose control in Chinese type 2 diabetic patients. To test this hypothesis, we plan to conduct this randomized controlled trial about low GI diet in Chinese diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese Type 2 diabetic patient.
2. Already performing self monitoring blood glucose ( SMBG ) with pre- and post-meal readings.
3. At least 50% of 2hr post-meal capillary blood glucose values are > 9 mmol/L.
4. A1c between 7.0 to 8.0% within 2 weeks of randomization.
5. Next follow-up is scheduled to at least 12 weeks or more if currently follow-up in TWEH.
6. On stable dose of anti-diabetic drug in the preceding 10 weeks.
7. No change in anti-DM drug in the next 10 week.
8. At least 18 years old.
9. Can read and understand consent form written in Chinese.
10. Can give informed consent.

Exclusion Criteria:

1. Unexplained hypoglycaemia in last 4 weeks.
2. Using rapid onset insulin ( such as Humalog, Novorapid, Actrapid HM, Mixtard HM, Novomix and Humalog Mix ).
3. Using acarbose.
4. Anaemia.
5. Known thalassaemia.
6. Suspected or confirmed iron deficiency.
7. On warfarin.
8. Renal impairment with serum creatinine > 150 umol/L
9. Active medical illness, such as hepatitis, malignancy, infection, inflammatory arthritis, etc.
10. Unable to follow low glycaemic index diet.
11. Currently participate in other study.
12. Mentally or cognitively disable.
13. Pregnant or lactating women.
14. Hospital Authority or TWEH staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood HbA1c | Baseline and week 10

SECONDARY OUTCOMES:
Change in pre- and 2-hour post-meal capillary blood glucose concentration | Baseline and week 10
Change in fasting blood glucose | Baseline and week 10
Change in lipid profile ( total cholesterol, triglycerides, LDL-C, HDL-C ) | Baseline and week 10
Change in blood ALT | Baseline and week 10
Change in body weight | Baseline and week 10
Change in blood pressure | Baseline and week 10

CONTACTS AND LOCATIONS:
Overall Officials: Ace Lee, MBBS, Principal Investigator — Department of Medicine and Rehabilitation, Tung Wah Eastern Hospital, Hospital Authority, Hong Kong
Locations (1):
- Tung Wah Eastern Hospital, Hospital Authority, Hong Kong SAR, Hong Kong SAR, China

REFERENCES:
- [Background] Brand-Miller J, Hayne S, Petocz P, Colagiuri S. Low-glycemic index diets in the management of diabetes: a meta-analysis of randomized controlled trials. Diabetes Care. 2003 Aug;26(8):2261-7. doi: 10.2337/diacare.26.8.2261. PMID 12882846
- [Background] Miller JB, Pang E, Bramall L. Rice: a high or low glycemic index food? Am J Clin Nutr. 1992 Dec;56(6):1034-6. doi: 10.1093/ajcn/56.6.1034. PMID 1442654
- [Background] Venn BS, Williams SM, Mann JI. Comparison of postprandial glycaemia in Asians and Caucasians. Diabet Med. 2010 Oct;27(10):1205-8. doi: 10.1111/j.1464-5491.2010.03069.x. PMID 20873364
- [Background] Jenkins DJ, Kendall CW, McKeown-Eyssen G, Josse RG, Silverberg J, Booth GL, Vidgen E, Josse AR, Nguyen TH, Corrigan S, Banach MS, Ares S, Mitchell S, Emam A, Augustin LS, Parker TL, Leiter LA. Effect of a low-glycemic index or a high-cereal fiber diet on type 2 diabetes: a randomized trial. JAMA. 2008 Dec 17;300(23):2742-53. doi: 10.1001/jama.2008.808. PMID 19088352